CLINICAL TRIAL: NCT04224519
Title: Consistency Study for Three Commercial Lots of Inactivated Poliomyelitis Vaccine Made From Sabin Strain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Collaborators: Yunnan Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20171217
Record Dates: First submitted 2020-01-06; First posted 2020-01-13 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Batch 1 of sIPV (Experimental): The first commercial batch of sIPV
  Interventions: Biological: sIPV batch 1
- Batch 2 of sIPV (Experimental): The second commercial batch of sIPV
  Interventions: Biological: sIPV batch 2
- Batch 3 of sIPV (Experimental): The third commercial batch of sIPV
  Interventions: Biological: sIPV batch 3

INTERVENTIONS:
Biological: sIPV batch 1 — Type I 30 DU, Type II 32 DU, Type III 45 DU
  Arms: Batch 1 of sIPV
Biological: sIPV batch 2 — Type I 30 DU, Type II 32 DU, Type III 45 DU
  Arms: Batch 2 of sIPV
Biological: sIPV batch 3 — Type I 30 DU, Type II 32 DU, Type III 45 DU
  Arms: Batch 3 of sIPV

SUMMARY:
A randomized and blind clinical consistency study for three commercial batches of Inactivated Poliomyelitis Vaccine Made From Sabin Strain (sIPV) for immunogenicity and safety evaluation.

DETAILED DESCRIPTION:
This randomized and blind clinical study includes three test groups with 400 infants for each group. Sample estimation for this study has been conducted using statistical methods.

A total of 1,200 2-month old healthy subjects were enrolled for inoculation of vaccine from 3 different lots with 1 month interval. All subjects received blood collection for immunogenicity test before and after primary immunization for evaluation of immunogenicity consistency, while safety observation was conducted within 30 days after each vaccination (30min via close safety monitoring, 0-7 days via participant diary card and 8-30 days via contact card for collection of adverse events) for safety evaluation of sIPV of 3 commercial lots.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants of 2 months of age
* The legal identity certificate (birth/household register) and vaccination certificate of the participants can be provided, and the legal guardian can provide the legal identity certificate (identity card).
* Guardians are able to understand the experimental vaccine, volunteer to participate in the study and sign informed consent for participation.
* Guardians are capable of using thermometer, graduated scale, filling diary card and contact card.
* Participants are not vaccinated with polio vaccine and immunoglobulin (except for Hepatitis b specific immunoglobulin) after birth, no vaccination of live vaccine within 28 days before enrollment and no vaccination of inactivated vaccine within 14 days before enrollment.
* Participants or guardians are able to obey and follow all study instructions, complete all the monitoring, and cooperate to complete collection of blood sample.
* Axillary temperature ≤37℃

Exclusion Criteria:

* Allergic to any active substance, inactive substance or materials used during production such as kanamycin.
* Patients with fever or acute disease.
* Have thrombocytopenia or hemorrhagic diseases
* Patients undergoing immunosuppressive therapy or immunodeficiency
* Have uncontrolled epilepsy or other progressive neurological disorders
* Other situations that the investigator consider as non-eligible

Ages: 2 Months to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-10-12 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate of neutralizing antibody | 1 month after primary immunization
  Blood samples were collected before and after immunization. Seroconversion rate of serum neutralizing antibody was determined. Intergroup differences analysis of the post-immunization positive conversion and ≥4-fold increase rate of antibody was performed.
Local and systemic adverse reactions | Within 1 month after primary immunization
  Safety monitoring for local and systemic adverse reaction within 30 days after 3-dose primary immunization via close monitoring or diary card.

SECONDARY OUTCOMES:
GMT of neutralizing antibody | 1 month after primary immunization
  Blood samples were taken before and after immunization for the determination of antibody level of serum neutralizing antibody. Intergroup differences analysis of antibody level was conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoqiang Liu, Principal Investigator — Disease prevention and control center of Yunnan province
Locations (1):
- Disease prevention and control center of Yunnan province, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No
Participants do not agree to share the individual data.

REFERENCES:
- [Derived] Yin Q, Zheng Y, Ying Z, Li J, Jiang Y, Bao W, Dou Y, Pu Y, Lei J, Yang H, Jiang R, Deng Y, Zhao Z, Pu J, Yang J, Li Y, Xu M, Cai W, Che Y, Shi L. Quantitative Analysis of the Instant and Persistent Inhibition Effects of Maternal Poliovirus Antibodies on the Immune Response in a Phase IV Trial of a Sabin Strain-Based Inactivated Poliovirus Vaccine. Vaccines (Basel). 2024 Feb 19;12(2):217. doi: 10.3390/vaccines12020217. PMID 38400200
- [Derived] Yin Q, Zheng Y, Ying Z, Li J, Jiang Y, Bao W, Dou Y, Pu Y, Lei J, Yang H, Jiang R, Deng Y, Zhao Z, Pu J, Yang J, Li Y, Xu M, Cai W, Che Y, Shi L. Immunogenicity and lot-to-lot consistency of booster shot with Sabin inactivated poliomyelitis vaccine in Chinese children aged 18-24 Months: A phase Ⅳ clinical trial. Vaccine. 2024 Mar 19;42(8):1973-1979. doi: 10.1016/j.vaccine.2024.02.042. Epub 2024 Feb 21. PMID 38388236
- [Derived] Jiang R, Liu X, Sun X, Wang J, Huang Z, Li C, Li Z, Zhou J, Pu Y, Ying Z, Yin Q, Zhao Z, Zhang L, Lei J, Bao W, Jiang Y, Dou Y, Li J, Yang H, Cai W, Deng Y, Che Y, Shi L, Sun M. Immunogenicity and safety of the inactivated poliomyelitis vaccine made from Sabin strains in a phase IV clinical trial for the vaccination of a large population. Vaccine. 2021 Mar 1;39(9):1463-1471. doi: 10.1016/j.vaccine.2021.01.027. Epub 2021 Jan 22. PMID 33487470